CLINICAL TRIAL: NCT02263235
Title: Use of Targeted Quantitative Proteomics and Metabolic Labelling With Stable Isotopes for the Diagnosis and the Investigation of Neurological Disorders and in Particular Alzheimer Disease
Brief Title: In Vivo Alzheimer Proteomics
Acronym: PROMARA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of the inclusion period
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Clermont-Ferrand (Other); International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 8652
Record Dates: First submitted 2014-09-18; First posted 2014-10-13 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Probable Alzheimer Disease; Parkinson Disease; Neurological Disease Without Cognitive Degradation; Brain Trauma; Acute Hydrocephaly
Keywords: Alzheimer disease (AD); diagnosis biomarkers; cerebrospinal fluid (CSF); targeted quantitative proteomics; mass spectrometry; stable isotope-labelled leucine
MeSH Terms: conditions — Parkinson Disease; Brain Injuries, Traumatic; Alzheimer Disease | interventions — Blood Specimen Collection; Urination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): 60 patients (20 probable AD, 20 Parkinson Disease (PK), 20 neurological disease without cognitive degradation)
  Interventions: Other: collection of CSF, blood, urine, saliva
- Group 2A (Experimental): 20 patients (patients with brain trauma, acute hydrocephaly), with temporary derivation of the CSF
  Interventions: Biological: administration of stable isotope-labelled leucine-
- Group 2B (Experimental): 30 patients (15 probable AD, 15 neurological disease without cognitive degradation)
  Interventions: Biological: administration of stable isotope-labelled leucine-

INTERVENTIONS:
Biological: administration of stable isotope-labelled leucine- — - administration of stable isotope-labelled leucine : by drip, for group 2A and group 2B. Group 1 (control group) : 1 collection of CSF. Group 2B : 4 collections of CSF, 24 hours after administration of stable isotope-labelled leucin. Group 2A (patients with brain trauma, acute hydrocephaly) : continuous collection of CSF, for 24 to 36 hours
  Arms: Group 2A; Group 2B
Other: collection of CSF, blood, urine, saliva — - administration of stable isotope-labelled leucine : by drip, for group 2A and group 2B. Group 1 (control group) : 1 collection of CSF. Group 2B : 4 collections of CSF, 24 hours after administration of stable isotope-labelled leucin. Group 2A (patients with brain trauma, acute hydrocephaly) : continuous collection of CSF, for 24 to 36 hours
  Arms: Group 1

SUMMARY:
In France, an estimated 860 000 patients are affected by Alzheimer Disease (AD) which represents, as in other developed countries, a major public health issue. In many cases, AD diagnosis is uncertain and its clinical evolution unpredictable. The exactitude of the diagnosis is however particularly important in the perspective of the validation and use of new therapeutic strategies in AD. Detection of cerebrospinal fluid (CSF) diagnosis biomarkers fell short in the detection, of atypical/mixed cases, of some differential diagnosis, and in differentiating rapid or slow clinical evolutions. Hence, CSF analysis gives a unique opportunity to detect and validate biomarkers in many neurological disorders. Nevertheless, in medical practice, CSF biological analysis is currently limited to a small number of analytes.Quantitative and targeted mass spectrometry, especially operated in the Multiple reaction monitoring mode (MRM), represents an alternative to immunodetection and could be used to detect specific biomarkers in complex matrices such as plasma by specifically discriminating the proteotypic peptides corresponding to each proteins. Mass spectrometry has also the ability to distinguish and quantify isotopically labelled and unlabeled selected targets. This ability was used in a publication by the group of R. Bateman (Washington University, St Louis, USA) who could, after administering stable isotope-labelled leucine, evaluate Ab synthesis and clearance in humans. This approach has an enormous potential to study the metabolism of proteins within the human CNS and consequently help in the understanding and diagnosis of neurological disorders.The main objective of this program is set up a targeted quantitative mass spectrometry method for existing and stable isotope-labelled CSF biomarkers in the neurological field; exploit this approach for diagnostic purpurses and to gain knowledge in the pathophysiology of diseases.

ELIGIBILITY:
Inclusion Criteria:

* Reports written consent, informed and signed by the patient and a trusted person
* Subject member or beneficiary of a social security system

Specific criteria for group 1 and 2B :

* Age between 55 and 85 years old for patients
* Subject with AD or other neurodegenerative disease (frontotemporal dementia, dementia with Lewy bodies, Parkinson disease)
* Subjects with chronic adult hydrocephalus (HCA) requiring depletion lumbar puncture (PL)

Specific criteria for group 2A :

- Adult patient requiring neurosurgery with CSF shunt (subject with brain trauma, acute hydrocephaly) and favorable evolution that allows removal of the shunt

Exclusion Criteria:

* Patient deprived of liberty by judicial or administrative decision
* Major protected by law
* Pregnancy, women of childbearing age with risk of pregnancy, or breast-feeding
* Presence of a transmissible viral disease (HlV, hepatitis B and C)
* Patient included in a clinical trial
* lnadequate cardiac, hepatic or severe renal disfunction
* Disease amino acid metabolism (Leucinose..)

Exclusion Criteria:

* Information clinical and para-clinical insufficient or unavailable
* Patient deprived of liberty by judicial or administrative decision
* Major protected by law
* Pregnancy, women of childbearing age with risk of pregnancy, or breast
* feeding
* Presence of a transmissible viral disease (HIV, hepatitis B and C)
* Patient included in a clinical trial
* Patient exclusion period relative to another protocol or for which the maximum annual compensation of 4500€ has been reached
* Inadequate cardiac, hepatic or severe renal
* Disease amino acid metabolism (Leucinose..)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-10-08 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
C13 Leucine incorporation in Amyloid peptides (1-40, 1-42) at different time points (in %) | 1.5 years
  Analysis of labelled samples with mass spectrometry. Data generated will be studied to validate the experimental model and understand the pathophysiology of neurological disorders. A collection of labelled biological samples will also be generated.
C13 Leucine incorporation in detectable peptides generated after trypsin digestion of biological fluids from patients (CSF, blood, urine, saliva) (in %) | 1.5 years
  C13 Leucine incorporation in detectable peptides generated after trypsin digestion of biological fluids from patients (CSF, blood, urine, saliva) (in %)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Lehmann, PU-PH, Principal Investigator — Laboratoire de Biochimie et Protéomique Clinique, IRMB St Eloi, CHRU de Montpellier
Locations (1):
- Laboratoire de Biochimie et Protéomique Clinique, CHU Montpellier, Montpellier, France